CLINICAL TRIAL: NCT03619993
Title: A Comparison of Pegfilgrastim (Neulasta®) Application Via Manual Injection Versus Injection Via an On-body Injector Regarding Patient Preference and Health Economics
Brief Title: Patient Preference for Pegfilgrastim (Neulasta®) Application Forms
Acronym: CONVENIENCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: iOMEDICO AG (Industry)
Collaborators: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IOM-040369
Record Dates: First submitted 2018-06-19; First posted 2018-08-08 (Actual); Last update posted 2019-12-17 (Actual); Status verified 2019-12

CONDITIONS: Non Hodgkin Lymphoma; Breast Cancer
Keywords: R-CHOP; G-CSF; Early breast cancer; Anthracycline/cyclophosphamide; 1st line; immunochemotherapy; taxane
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A: Start with On-body injector (Experimental): 4 consecutive cycles of treatment in total, with 2 cycles of treatment with pegfilgrastim pre-filled syringe (PS) and 2 cycles of treatment with On-body injector (OBI) for pegfilgrastim in an alternating sequence (OBI-PS-OBI-PS)
  Interventions: Device: On-body injector; Device: Pre-filled syringe
- Arm B: Start with pre-filled syringe (Experimental): 4 consecutive cycles of treatment in total, with 2 cycles of treatment with pegfilgrastim pre-filled syringe (PS) and 2 cycles of treatment with On-body injector (OBI) for pegfilgrastim in an alternating sequence (PS-OBI-PS-OBI)
  Interventions: Device: On-body injector; Device: Pre-filled syringe

INTERVENTIONS:
Device: On-body injector — Medical device for subcutaneous injection of a supportive medicine (Pegfilgrastim) automatically after 27 hours after application of device.
Device: Pre-filled syringe — For subcutaneous injection of a supportive medicine (Pegfilgrastim).

SUMMARY:
The study aims to compare two application forms (pre-filled syringe and On-body injector) of the same active drug (pegfilgrastim) in adult patients under chemotherapy regarding patient preference and health economics. Chemotherapy will be supported with pegfilgrastim for four subsequent chemotherapy cycles using alternating application forms.

DETAILED DESCRIPTION:
Neutropenia is one of the most common side effects of myelosuppressive chemotherapy. Febrile neutropenia and infectious complications are associated with chemotherapy dose delays and reductions and an increased risk of hospitalization. Prophylaxis with recombinant G-CSFs reduces the incidence, severity and duration of CIN and the risk of developing FN. Pegfilgrastim is available for over 10 years and is specified in the SmPC to be applied at least 24 hours after cytotoxic chemotherapy. For this application patients often have to return to their physician one day after chemotherapy treatment for the sole purpose of receiving pegfilgrastim subcutaneous (s.c.) injection. For different reasons, some of the patients requiring pegfilgrastim may not be able to return at this day and thus may not receive pegfilgrastim in accordance with the SmPC. The On-body injector for pegfilgrastim provides an option for patients not to return to the clinic/medical office the day after chemotherapy for their pegfilgrastim injection. The kit includes a single-use prefilled syringe co-packed with the On-body injector for pegfilgrastim. The On-body injector is applied to the patient's skin at the day of chemotherapy treatment and it automatically delivers pegfilgrastim approximately 27 h after the On-body injector was applied to the patient's skin.

Patient-reported outcomes on preference for either application form can help to guide physicians' treatment choice, particularly in terms of application of the same active substance, in this study pegfilgrastim.

This study aims to compare the two application forms of pegfilgrastim (pegfilgrastim pre-filled syringe vs. On-body injector for pegfilgrastim) with regard to patient preference and health economy. A trial design with randomization of patients to receive the two application forms of pegfilgrastim in an alternating sequence for 4 cycles starting with either On-body injector for pegfilgrastim (Arm A) or pegfilgrastim pre-filled syringe (Arm B) was chosen. In this way, all patients will receive both application forms in order to be able to decide for their individual preference. Four cycles (that means each patient will receive each application form of pegfilgrastim twice) should be a sufficient number for the patient to make a decision. This design with two treatment arms serves to exclude a systematic bias that might be generated when starting with the same application form for all patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients with early breast cancer planned to receive 3 weekly or dose-dense anthracycline/cyclophosphamide combination or 3 weekly taxane containing chemotherapy regimen or patients with NHL planned to receive R-CHOP-14 or R-CHOP-21 immunochemotherapy as 1st-line treatment with the indication for G-CSF prophylaxis with pegfilgrastim for the prevention of FN and reduction in CIN duration. Patients have to be included before start of their (immuno-) chemotherapy.
* ECOG (Eastern Cooperative Oncology Group) performance status 0, 1 or 2
* Life expectancy > 3 months
* Absolute neutrophil count ≥ 1.5 x 109/L
* Ability to read and understand German
* Signed informed consent

Exclusion Criteria:

* Hypersensitivity to the active substance or to any of the excipients
* Subject is currently enrolled or has not yet completed at least 30 days since ending other investigational device or drug trial(s) or is receiving investigational agent(s)
* Active infection or any serious underlying medical condition, which would impair the ability of the patient to receive protocol treatment
* Prior bone marrow or stem cell transplantion
* Subject of child-bearing potential is evidently pregnant (e.g. positive HCG (Human Chorionic Gonadotropin) test) or is breast feeding
* Subject is not using adequate contraceptive precautions.
* Other conditions which, in the opinion of the investigator, make participation in an investigational trial of this nature a poor risk
* Concerns for subject's compliance with the protocol procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 404 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-09-10 (Actual); Study Completion 2019-09-10 (Actual)

PRIMARY OUTCOMES:
Patient preference for type of pegfilgrastim application assessed via project specific survey answered after 4 applications. | 4 cycles of chemotherapy, i.e. 8 to 12 weeks (depending on chemotherapeutic regimen)
  Percentage of patients favoring pegfilgrastim application via On-body injector. Patients are answering the questionnaire after 4 applications of pegfilgrastim in total, with On-body injector and pre-filled syringes used in alternating sequence (each type of application administered two times in total).

SECONDARY OUTCOMES:
Time point of pegfilgrastim application within a chemotherapy cycle | 4 cycles of chemotherapy, i.e. 8 to 12 weeks (depending on chemotherapeutic regimen)
  The number of hours between chemotherapy application and pegfilgrastim application in each of the 4 observed chemotherapy cycles.
Patient preference for pegfilgrastim application assessed via project specific survey answered at time of enrollment | at enrollment
  Percentage of patients favoring pegfilgrastim application via On-body injector. Patients are answering the questionnaire before initial application.
Impact of type of pegfilgrastim application on daily life of the patient assessed by direct questioning using project specific patient survey. | 4 cycles of chemotherapy, i.e. 8 to 12 weeks (depending on chemotherapeutic regimen)
  Percentage of patients reporting a certain impact level with respect to the type of pegfilgrastim application. Patient questionnaires will be answered after pegfilgrastim application in each of the 4 observed chemotherapy cycles.
Percentage of nurses favoring pegfilgrastim application via On-body injector at study start and at end of study as stated via a project specific nurse survey | from first enrollment to end of study of last patient at a site (= end of cycle 4 of last patient, expected to be latest 2.5 years after study start)
  Percentage of nurses favoring pegfilgrastim application via On-body injector. Nurses are answering the questionnaire at study start and at the end of the study.
Preference of investigators for either type of pegfilgrastim application at study start und at end of study assessed via project specific investigator survey | from first enrollment to end of study of last patient at a site (= end of cycle 4 of last patient, expected to be latest 2.5 years after study start)
  Percentage of investigators favoring pegfilgrastim application via On-body injector. Investigators are answering the questionnaire at study start and at the end of the study.
Cost factors for the health care system for both types of application of pegfilgrastim | 4 cycles of chemotherapy, i.e. 8 to 12 weeks (depending on chemotherapeutic regimen)
  Cost factors are assessed via project specific patient survey addressing time, travel expenses and support needed to receive pegfilgrastim application.

OTHER OUTCOMES:
Resource utilization at site for either type of application assessed via project specific study nurse survey | at end of study of last patient at a site (= end of cycle 4 of last patient, expected to be latest 2.5 years after study start)
  Resource utilization at site is assessed via study nurse questionnaire addressing involvement of site staff and further site resources to apply pegfilgrastim.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Metz, Dr. med., Study Chair — OSP Göttingen - Gemeinschaftspraxis Dres. Meyer, Ammon, Metz und Müller
Locations (47):
- Germany (47):
  - Research Site, Aschaffenburg
  - Research Site, Augsburg
  - Research Site, Berlin
  - Research Site, Bonn
  - Research Site, Celle
  - Research Site, Dresden
  - Research Site, Erfurt
  - Research Site, Flensburg
  - Research Site, Frankfurt (Oder)
  - Research Site, Freiburg im Breisgau
  - Research Site, Georgsmarienhütte
  - Research Site, Goslar
  - Research Site, Göttingen
  - Research Site, Halberstadt
  - Research Site, Halle
  - Research Site, Hanover
  - Research Site, Heidelberg
  - Research Site, Herne
  - Research Site, Hildburghausen
  - Research Site, Hildesheim
  - Research Site, Kaiserslautern
  - Research Site, Kassel
  - Research Site, Köthen
  - Research Site, Krefeld
  - Research Site, Mannheim
  - Research Site, Mayen
  - Research Site, Moers
  - Research Site, Mühlhausen
  - Research Site, Mülheim
  - Research Site, München
  - Research Site, Naunhof
  - Research Site, Neunkirchen
  - Research Site, Neustadt in Sachsen
  - Research Site, Nordhorn
  - Research Site, Offenbach
  - Research Site, Oldenburg
  - Research Site, Ostfildern
  - Research Site, Passau
  - Research Site, Plauen
  - Research Site, Ratingen
  - Research Site, Rostock
  - Research Site, Singen
  - Research Site, Sömmerda
  - Research Site, Spremberg
  - Research Site, Stolberg
  - Research Site, Stralsund
  - Research Site, Würselen

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Metz M, Semsek D, Rogmans G, Hutzschenreuter U, Fietz T, Harde J, Zacharias S, Hielscher C, Lorenz A, Zahn MO, Guth D, Liebers S, Berghorn M, Grebhardt S, Matillon CD, Egerer G, Potthoff K. Patient, nurse, and physician preferences: final results of the CONVENIENCE study evaluating pegfilgrastim prophylaxis via pre-filled syringe or on-body injector in cancer patients. Support Care Cancer. 2021 Nov;29(11):6633-6643. doi: 10.1007/s00520-021-06230-9. Epub 2021 May 6. PMID 33956213